CLINICAL TRIAL: NCT05692232
Title: The Efficacy of Manual Therapy and Pressure Biofeedback Guided Deep Cervical Flexor Muscle Strength Training on Pain and Functional Limitations in Individuals With Cervicogenic Headaches. A Randomized Comparative Study
Brief Title: The Efficacy of Manual Therapy and Pressure Biofeedback Guided Strength Training on Pain and Functional Limitations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Majmaah University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2022-04
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Cervicogenic Headache
Keywords: Pressure biofeedback; Deep cervical flexor muscles; Muscle Strengthening; Manual therapy; Pain; Disability
MeSH Terms: conditions — Post-Traumatic Headache; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Thirty participants randomly allocated to group 1. All the participants received a pressure biofeedback guided deep cervical flexor muscle strength training along wth conventional intervention.
  Interventions: Other: Pressure biofeedback guided DCFM strength training; Other: Conventional intervention
- Group 2 (Active Comparator): Thirty participants randomly allocated to group 2. All the participants received a manual therapy along wth conventional intervention.
  Interventions: Other: Manual therapy; Other: Conventional intervention

INTERVENTIONS:
Other: Pressure biofeedback guided DCFM strength training — A pressure biofeedback guided DCFM strength training was carried out according to the Jull protocol. Keeping the participant's cervical spine in a neutral position and ensuring a stabilizer pressure biofeedback unit placed beneath the cervical lordosis. The pressure sensor was inflated at 20mm Hg. The participants were asked to nod their heads slowly. As the DCFM is activated, the cervical lordosis gently flattens, and the pressure sensor measures an increase in pressure. The activation score is the maximum pressure that can maintain for 10 seconds.
  Arms: Group 1
Other: Manual therapy — A manual therapy, including a slow, sustained elongation of muscles with a holding period of 7-10 seconds and a superficial oscillatory mobilization (grade-I) with 1-2 oscillations per second for 30 seconds per session was performed on the DCFM and at the cervical spine (C0-C5), respectively. The participants were asked to lie supine and prone while delivering stretching and mobilization, respectively.
  Arms: Group 2
Other: Conventional intervention — A hot pads was applied for 20minutes underneath the cervical spine covering either side of shoulder in a relaxed supine position.

SUMMARY:
Cervicogenic headache (CGH) is a widespread illness that results in excruciating pain and a sizable functional handicap. Deep cervical flexor muscle (DCFM) strength and endurance were also worse in CGH patients. This study aimed to determine the efficacy of manual therapy and pressure biofeedback-guided DCFM strength training on pain intensity and functional limitations in individuals with CGH.

DETAILED DESCRIPTION:
The study followed a two-arms parallel group randomized comparative design, including sixty individuals with CGH, and they were allocated into two groups at random. For three consecutive weeks, in addition to the conventional treatment common to both groups, groups 1 and 2 received pressure biofeedback-guided DCFM strength training and manual therapy, respectively. At baseline, the first week, the second week, and the third week post intervention, pain intensity and functional limitations were evaluated using the visual analog scale (VAS), the number of headache days per week, and the headache disability inventory (HDI) questionnaire. The main effects of the intervention were evaluated for a between-group factor, within-group factor, and interaction between time and groups over/at multiple time points. Data was analyzed using an independent t-test, mixed design 2-way ANOVA, with keeping the level of significance 'p' at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individual with a diagnosed case of cervicogenic headache with unilateral head pain without side shift or bilateral head pain with a dominant side that hurts more than the other side, sustained awkward head positioning, external pressure over the upper cervical or occipital region on the symptomatic side.
* Aged between 25 and 50 years
* Patients with recurrent CGH and chronic mechanical neck discomfort that has persisted for longer than three months.
* A positive cervical flexion rotation test.

Exclusion Criteria:

* a negative cervical flexion rotation test.
* Subjects had a history of any of the following conditions: a fractured vertebral column or previous surgery on it; spinal stenosis; a prolapsed disc; temporomandibular joint dysfunction or headaches involving the autonomic nervous system; vertigo or visual disturbance; or a congenital condition of the cervical spine.
* Showed non-cooperation

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 6 weeks
  The pain intensity was assessed by a visual analogue scale. It is a reliable and valid tool to measure the pain intensity. It is an objective line marked with zero indicate no pain and ten indicate maximum unbearable pain at the either end of the line. Individuals are asked to show the level of pain by putting their fingers on the line between either ends.
Functional limitations | 6 weeks
  The functional limitation due to cervicogenic headache was evaluated by a self-rated questionnaire called as, Headache Disability Index. A minimum and maximum scores ranges from 0 to 100. a score of 10-28 is considered to constitute mild disability; 30-48 is moderate disability; 50-68 is severe disability; 72 or more is complete disability.

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT, Principal Investigator — King Saud University
Locations (1):
- Department of Rehabilitation Sciences, College of applied Medical Science, King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasan S, Bharti N, Alghadir AH, Iqbal A, Shahzad N, Ibrahim AR. The Efficacy of Manual Therapy and Pressure Biofeedback-Guided Deep Cervical Flexor Muscle Strength Training on Pain and Functional Limitations in Individuals with Cervicogenic Headaches: A Randomized Comparative Study. Pain Res Manag. 2023 Aug 14;2023:1799005. doi: 10.1155/2023/1799005. eCollection 2023. PMID 37608909